CLINICAL TRIAL: NCT01936129
Title: Investigating the Neuroprotective Effect of Cop-1 in Acute Primary Angle Closure
Brief Title: Investigating the Neuroprotective Effect of Cop-1 (Copaxone) in Acute Primary Angle Closure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Prof Aung Tin, Professor, Singapore Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R624/45/2008
Record Dates: First submitted 2013-08-28; First posted 2013-09-05 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma, Angle-closure, Primary, Acute
MeSH Terms: conditions — Glaucoma | interventions — Glatiramer Acetate; Coat Protein Complex I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Copaxone (Active Comparator): COPAXONE (glatiramer acetate) will be administered as a subcutaneous dose (20mg) once, one injection no later than 7 days from the initiation of the attack, and 1 more injection administered one week after the first injection.
  Interventions: Drug: Copaxone
- Placebo (Placebo Comparator): Placebo (buffered normal saline w/v)will be administered as a subcutaneous dose, one injection no later than 7 days from the initiation of the attack, and 1 more injection administered one week after the first injection.
  Interventions: Drug: Placebo (buffered normal saline w/v)

INTERVENTIONS:
Drug: Copaxone
  Other Names: Cop 1; glatiramer acetate
  Arms: Copaxone
Drug: Placebo (buffered normal saline w/v)
  Arms: Placebo

SUMMARY:
This is a randomised controlled trial to assess the neuroprotective effect of Cop-1 (Copaxone) in patients with acute primary angle closure (APAC). The standardized management of APAC will include medical therapy to reduce intraocular pressure (IOP), followed by laser peripheral iridotomy. Cop-1 will be administered in addition to standard therapy as a subcutaneous dose once within 24 hours of presentation, and then one week later (total 2 injections). The control group will have placebo in addition to standard regimen. Subjects in the study will have visual field test performed with the Humphrey Visual Field Analyzer II, retinal nerve fibre layer (RNFL) thickness measured with the Stratus optical coherence tomography (OCT) and Optic nerve head evaluated with the Heidelberg retinal tomography (HRT). At least 2 baseline visual field tests will also be performed in the first week. Subsequent visits will be at week 4, 8, 12 and 16. The outcome criteria will be difference in visual field, RNFL thickness, and optic nerve head structural changes.

DETAILED DESCRIPTION:
Aim To assess the neuroprotective effect of Cop-1 (Copaxone) in reducing functional and structural damage after acute primary angle closure (APAC)

Outcome measures:

The primary outcome measures will be the point-wise linear regression in the visual fields.

The secondary outcome measure will be the evaluation of structural changes, namely, RNFL thickness and Optic disc changes as measured by stratus OCT and HRT respectively.

Study population

The study population (n=196; 1:1 randomisation) will be patients with APAC attending the Singapore National Eye Centre who fulfil the inclusion criteria and are willing to take part in the study.

Study design:

The study design is a randomized, placebo controlled, double blinded trial where patients with APAC will be randomized to receive either Cop-1 (Copaxone) or placebo in addition to the standard medical therapy.

An interim analysis will be conducted after 40 patients complete the trial. Routine examination will be done at all visits.

ELIGIBILITY:
Inclusion Criteria:

* • patients with APAC who present to the centre not later than 7 days from the initiation of the attack.

  * the presence of at least two of the following symptoms: ocular or periocular pain, nausea or vomiting or both, and an antecedent history of blurring of vision with haloes;
  * a presenting intraocular pressure of at least 28 mm Hg on Goldmann applanation tonometry;
  * the presence of at least three of the following signs: conjunctival injection, corneal epithelial oedema, middilated unreactive pupil, and shallow anterior chamber;
  * the presence of an occludable angle in the affected eye on gonioscopy;
  * Age more than 21 years.
  * Informed consent

Exclusion Criteria:

* • evidence of a prior acute angle closure attack (the presence of iris whorling, focal iris atrophy, or glaucomflecken with a history of an acute red eye and decreased vision). This will not include senile iris and sphincter atrophy);

  * Pre-existing chronic angle closure glaucoma in the eye with APAC
  * secondary causes of angle closure like subluxed lens, uveitis, trauma and neovascular glaucoma;
  * cataract that is deemed significant enough to require surgery during the course of the trial or that makes field testing or optic disc imaging not technically possible- visual acuity less than 6/36 due to any type of cataract;
  * corneal abnormalities, media opacities, or retinal abnormalities that would affect scanning laser polarimetry;
  * previous intraocular surgery;
  * currently pregnant or nursing women, or women considering pregnancy;
  * Severe health problems precluding follow-up such as end-stage heart disease, kidney disease, respiratory disease, or cancer and life expectancy less than one year.
  * History of allergy to mannitol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Visual field progression using point-wise linear regression. | 16 weeks

SECONDARY OUTCOMES:
The secondary outcome measure will be the evaluation of structural changes of the optic nerve head. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tin Aung, FRCOphth,PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore, Singapore